CLINICAL TRIAL: NCT05908409
Title: A Phase 1/2 Multicenter, Open-label, Dose-escalation Study of IDP-121 in Patients With Relapsed/Refractory Hematologic Malignancies (CASSANDRA)
Brief Title: A Phase 1/2 Study of IDP-121 in Patients With Relapsed/Refractory Hematologic Malignancies
Acronym: CASSANDRA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: IDP Discovery Pharma S.L. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IDP-121-1
Record Dates: First submitted 2023-05-03; First posted 2023-06-18 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma (MM); Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Double Hit Lymphoma; High Grade B-Cell Lymphoma, Not Otherwise Specified; Chronic Lymphocytic Leukemia (CLL); Triple Hit Lymphoma
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Large B-Cell, Diffuse; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation: IDP-121 0.015 Up to 0.70 mg/kg (Experimental): IDP-121 will be administered as a 4-hours i.v. infusion twice a week (3 weeks on, 1 week off) on days 1, 4, 8, 11, 15 and 18 in 28-day treatment (a Cycle) (Table 4). A minimum interval of 3 days and no more than 5 days between dosing is allowed.
  Patients can receive IDP-121 until disease progression, unacceptable toxicity or any other discontinuation criteria are met, or for a maximum treatment period of 1 year, whichever occurs first. Patients at the RP2D may enter the expansion phase.
  Interventions: Drug: IDP-121
- Expansion Phase: IDP-121 at RP2D (Experimental): Additional 17 patients will be enrolled for treatment at the RP2D level to further study safety and evaluate efficacy. DP-121 will be administered as a 4-hours i.v. infusion twice a week (3 weeks on, 1 week off) on days 1, 4, 8, 11, 15 and 18 in 28-day treatment Patients can receive IDP-121 until disease progression, unacceptable toxicity or any other discontinuation criteria are met, or for a maximum treatment period of 1 year, whichever occurs first.
  Interventions: Drug: IDP-121

INTERVENTIONS:
Drug: IDP-121 — IDP-121 is a new chemical entity specifically designed to directly target cMyc protein that has demonstrated activity in multiple liquid and solid tumor cell lines and preclinical animal models

SUMMARY:
The main aims of this 2-part study are:

* Phase I: To determine the maximum tolerated dose (MTD) and the recommended phase 2 dose (RP2D) of IDP-121 in patients with multiple myeloma (MM), diffuse large B cell lymphoma not otherwise specified (DLBCL-NOS), high-grade B cell lymphoma with double or triple hit rearrangement (HGBL-DH/TH) and HGBL-NOS, and chronic lymphocytic leukemia (CLL).
* Phase II: To evaluate the overall response rate (ORR), duration of response (DoR), time to progression (TTP), progression-free survival (PFS), event-free survival (EFS) and Overall survival (OS), in patients with MM, DLBCL-NOS, HGBL-DH/TH, HGBL-NOS or CLL treated with IDP-121 at the recommended Phase 2 Dose (RP2D).

DETAILED DESCRIPTION:
This study is an open-label, multicenter, Phase 1/2 study with a Dose-Escalation phase (Phase 1) and an Expansion phase (Phase 2).

Dose-Escalation (Phase 1): The dose-escalation phase will follow a classical 3+3 design but the first patient (sentinel) will be treated at dose level 1 (0.015 mg/kg) for one cycle, and, if no Dose-Limiting Toxicities (DLTs) occur, at dose level 2 (0.032 mg/kg) from cycle 2 onwards. Once the patient 1 (sentinel) is allowed to enter dose level 2, two additional patients will be enrolled to complete the cohort at dose level 2, and the dose-escalation phase will continue the 3+3 design. DLTs will be assessed based on the safety observed in cycle 1 (28 days) for all patients except for patient 1 (sentinel) where DLT will be assessed on safety observed in cycle 1 (at dose level 1) and cycle 2 (at dose level 2). For the first trial patient (sentinel) a single cycle will be completed (28 days) at dose level 0.015 mg/kg. Doses will not be escalated before all patients entered at the current dose level have been treated and observed for at least one complete cycle (28 days) at the intended dose- cohort IDP-121 dose and the number of DLTs among those patients in their first cycle has been determined. Before each escalation, Clinical Investigators will be consulted as part of a cohort review meeting to review and discuss all data (including safety, PK, PD and efficacy data) and agree on a dose-escalation, as appropriate.

During the study, the Sponsor and Investigators may request that cohorts be enlarged or that intermediate doses between 2 planned escalation steps be explored based on all data existing at that time, including emerging safety and efficacy data and determinations of PK and PD. Also, the study will allow for alternative IDP-121 doses and/or schedules to be evaluated based on emerging data e.g., once a week dosing of IDP-121 (instead of twice a week). Data from all patients at all dose levels will be used to guide further dose-escalation or/and the MTD/RP2D.

Expansion-Phase (Phase 2): Additional 17 patients will be enrolled for treatment at the RP2D level to further study safety and evaluate efficacy. Patients will receive 28-day cycles up to a maximum of 12 cycles of treatment or until any IDP-121 treatment discontinuation criteria are met (disease progression, unacceptable toxicity, etc). Patients in the Expansion- Phase may include one or more tumor types from those evaluated in dose-escalation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Performance status (ECOG) ≤ 2
3. Life expectancy ≥3 months
4. Patient is, in the investigator's opinion, willing and able to comply with the protocol requirements.
5. Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
6. Patients diagnosed with chronic lymphocytic leukemia (CLL), B-cell lymphomas, and multiple myeloma (MM) who are ineligible to reveive the available treatments.
7. Adequate hematological or biochemical parameters as specified below

   1. Hemoglobin > 8.0 g/dl (without transfusion support within 7 days)
   2. Platelets count > 75 x109/L (without transfusional support within 7 days). In patients with bone marrow infiltration, the platelets count may be ≥50 x109/L.
   3. Absolute neutrophil count (ANC) > 0.75 x109/L (without G-CSF support within 7 days)
   4. Aspartate transaminase (AST): <2.5 x the upper limit range (in patients with no liver metastases or <5 x ULN in patients with liver metastases)
   5. Alanine transaminase (ALT): < 2.5 x the upper limit range (in patients with no liver metastases or <5 x ULN in patients with liver metastases)
   6. Total bilirubin: < 2 x the upper limit range.
   7. Calculated or measured creatinine clearance: >30 mL/min (calculated from the Cockcroft-Gault formula).
8. Left ventricular ejection fraction > 50% or above the Institutional Lower Limit of Normal (LLN), whichever is lower, determined by echocardiogram.

Exclusion Criteria:

1. Persistent clinically significant non-hematological toxicity related to previous treatments. The presence of alopecia and NCI-CTC grade <2 symptomatic peripheral neuropathy is allowed.
2. Pregnant or lactating women; men and women of reproductive potential* (as defined in the Appendix 2) who are not using effective contraceptive methods (combined hormonal contraception associated with inhibition of ovulation; progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomised partner, sexual abstinenence).

   *A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. A man is considered fertile after puberty unless permanently sterile by bilateral orchidectomy.
3. History of any other neoplastic disease in the last five years (except basal cell carcinoma, skin epithelioma or carcinoma in situ of any site)
4. History of clinically significant hypotension.
5. History of clinically significant allergic or hyper-sensitivity reactions.
6. History or known clinically significant vascular disease or known high risk of vascular disease (as assessed by the treating physician) including (but not limited to):

   * Thromboembolism
   * Peripheral arterial disease
   * Vasculitis
7. Other relevant diseases or adverse clinical conditions:

   * Congestive heart failure or angina pectoris, myocardial infarction within 12 months before inclusion in the study.
   * Uncontrolled arterial hypertension or cardiac arrhythmias (i.e., requiring a change in medication within the last 3 months or hospital admission within the past 6 months).
   * History of significant neurological or psychiatric disorders
8. Clinically significant or active infection.
9. Significant non-neoplastic liver disease (e.g., cirrhosis, active chronic hepatitis)
10. The patient is known to be human immunodeficiency virus (HIV) positive, unless the patient is on antiviral therapy with HIV RNA levels <50 copies/mL; Hepatitis B surface antigen-positive or active hepatitis C infection, unless treated with undetectable hepatitis B DNA or hepatitis C RNA levels; or active CMV infection (IgM positive).
11. Concomitant anti-tumor therapy within 14 days prior to Day 1 of Cycle 1.
12. Prior allogeneic transplantation in the last 3 months or currently active GVHD with immunosuppressive treatment
13. Limitation of the patient's ability to comply with the treatment or follow-up protocol.
14. If a COVID-19 vaccine is administered, it should be done >72 hours prior to study treatment initiation or after the completion of the dose-limiting toxicity (DLT) period (if patient is participating in the dose-escalation phase").

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2026-03-22 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Dose Escalation | Through 1 treatment cycle (each cycle is 28 days)
  Maximum tolerated dose (MTD)
Phase 1: Dose Escalation | Through 12 treatment cycles (each cylce is 28 days) or until End of Treatment, whatever occurs first
  Recommended phase 2 dose (RP2D)
Phase 2: Expansion Phase | Based on iwCLL 20181, IMWG 20162, and the Lugano 20143 criteria for CLL, MM and Lymphomas, respectively; assessed at the end of study (12 months)
  Overall Response Rate (ORR)

SECONDARY OUTCOMES:
Phase 2: Expansion Phase | From disease response to disease progression, up to 12 months
  Duration of response (DoR)
Phase 2: Expansion Phase | From the first treatment day to day of the objective disease progression through study completion, an average of 12 months
  Time to progression (TTP)
Phase 2: Expansion Phase | From first treatment day to the first sign of disease progression or death from any cause assessed up to 12 months.
  Progression-free survival (PFS)
Phase 2: Expansion Phase | From first treatment day to disease progression, death, or discontinuation of treatment from any cause through study completion, an average of 12 months
  Event-free survival (EFS)
Phase 2: Expansion Phase | From first treatment day to death from any cause, up to 12 months
  Overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Ocio San Miguel, MD, PhD, Principal Investigator — Hospital Universitario Marqués de Valdecilla
Locations (11):
- Spain (11):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario de Salamanca, Salamanca, Castille and León
  - Hospital Universitari Vall d'hebron, Barcelona
  - Hospital Durán i Reynals - ICO L´Hospitalet, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital de Clinico Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor´s web page — https://www.idp-pharma.com/